CLINICAL TRIAL: NCT01108042
Title: Phase I/II Study of Split-dose TPF-Induction Chemotherapy Before Surgery of Oropharyngeal and Cavity of the Mouth Cancer
Brief Title: TPF-Induction Chemotherapy of Oropharyngeal and Cavity of the Mouth Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orlando Guntinas-Lichius, Prof. Dr. med. (Other)
Responsible Party: Sponsor-Investigator, Orlando Guntinas-Lichius, Prof. Dr. med., Professor Dr. med., University of Jena
Organization: University of Jena (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TISOC-1; 2009-011902-41 (EudraCT Number)
Record Dates: First submitted 2010-04-14; First posted 2010-04-21 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Oropharynx Cancer; Squamous Cell Carcinoma of the Oral Cavity
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Taxotere, Cisplatin, 5-Fluorouracil (5-FU) (Experimental): Phase 1: Intravenous infusion of 40 mg/m² Taxotere and 40 mg/m² Cisplatin followed by 24 h-infusion of 2000 mg/m² 5-FU on day 1 and day 8 every 3 weeks. If possible an escalation to 50 mg/m² Taxotere and 50 mg/m² Cisplatin can be carried out.
  Interventions: Drug: Taxotere, Cisplatin, 5-Fluorouracil (5-FU)

INTERVENTIONS:
Drug: Taxotere, Cisplatin, 5-Fluorouracil (5-FU) — Phase 1: Intravenous infusion of 40 mg/m² Taxotere and 40 mg/m² Cisplatin followed by 24 h-infusion of 2000 mg/m² 5-FU on day 1 and day 8 every 3 weeks. If possible an escalation to 50 mg/m² Taxotere and 50 mg/m² Cisplatin can be carried out. Phase 2: Optimal dose of phase 1 will be given.
  Other Names: Docetaxel

SUMMARY:
A combination therapy of Docetaxel, Cisplatin und 5-Fluorouracil (= TPF) will be used in patients with resectable oropharyngeal and cavity of the mouth cancer. To improve the compatibility of the TPF-induction without decreasing the efficacy the dose will be given on day 1 and 8 instead of applying the whole dose on day 1 every 3 weeks.

In the phase I-part of the trial the optimal therapeutic dose of Docetaxel and Cisplatin will be defined.

In the phase II-part the progression-free survival after 2 years will be assessed in patients treated with the optimal therapeutic dose.

DETAILED DESCRIPTION:
Local advanced Oropharyngeal and cavity of the mouth Cancer are often treated with a combination of surgery and/or radiation and /or chemotherapy.

Despite of therapy improvement there are only little advances in progression-free survival and overall survival.

Therefore new therapy concepts are needed. The advantage of the induction chemotherapy is the possibility of tumor response assessment during chemotherapy and may present a selection criterion for organ preservation.

In order to minimize the time between chemotherapy and surgery it is important to have an early answer for the tumor response. In this study response will be assessed after the first cycle of chemotherapy. Patients showing no tumor response will be operated at once. The other patients will receive further cycles of chemotherapy.

Toxicity of the induction chemotherapy have to be moderate because surgery should not be delayed.

To improve the tolerance of induction therapy the medication dose isn't given on day 1 every 3 weeks, but is dispersed on day 1 and day 8, q3weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histological proven, resectable squamous epithelial carcinoma of the oropharynx and the cavity of the mouth
2. R0-resection possible
3. All T N2 M0 / all T N3 M0 / if T3 or T4a also N0-1 M0
4. Leucocytes > 4000/mm³ bzw. neutrophils > 2000/mm³, thrombocytes > 100000/mm³
5. adequate kidney function, defined as serum creatinine und urea in normal range, Creatinine clearance > 60 ml/min
6. adequate liver function with glutamate oxaloacetate transaminase (SGOT), glutamate pyruvate transaminase (SGPT) and bilirubin in normal range
7. electrolytes in normal range
8. risks of anesthesia complications normal or minor increased
9. Eastern Cooperative Oncology Group (ECOG) 0-2 / Karnofsky >= 60%
10. Age 18 - 80 years
11. signed written informed consent
12. effective contraception for both male and female subjects if the risk of conception exists

    Exclusion Criteria:
13. T1 N0 M0 / T1 N1 M0 / T2 N0 M0 / T2 N1 M0
14. Resection without curative intention: primary tumor is not treatable with resection methods
15. Infiltration of the lower jaw
16. M1 status
17. Tumor not measurable with Innovation Center Computer Assisted Surgery (ICCAS) methods
18. No prior chemotherapy or radiation (a primary surgery is allowed)
19. Metachronous or oder synchronous malignoma (Exception: basal cell carcinoma)
20. Life expectance < 3 months
21. ECOG > 2; Karnofsky < 60%
22. acute infections or fever
23. known HIV-infection or other immune suppression
24. severe cardio pulmonary concomitant diseases
25. chronic disease with continuous therapy (uncontrolled diabetes, rheumatoid arthritis) especially continuous therapy with steroids
26. other concomitant diseases which, in the investigator's opinion, would exclude the patient from the study
27. Contraindications which permit a therapy with Docetaxel, Cisplatin, 5-FU or radiation therapy
28. missing patient's compliance
29. regular Follow-up visits not possible
30. Pregnancy or lactation period
31. legal incapacity or limited legal capacity
32. Participation in another clinical trial or administration of a not approved substance within 30 days before registration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-11; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Determination of progression-free survival after 2 years | 24 months

SECONDARY OUTCOMES:
Overall survival after 2 years | after 2 years
Determination of the efficacy of the induction therapy | after 1, 12 and 24 months
  CT or magnetic resonance tomography (MRT) of the neck region
Function of swallowing according the penetration-aspiration-scale | 0,1, 6, 12, 18, 24 months
  assessed according the penetration-aspiration-scale (PAS, Rosenbek et al. 1996) and according measuring after Prosiegel (Prosiegel et al. 2002).
Adverse events as a measure of safety and tolerability | once a week
  The number of patients with adverse events will be evaluated. Adverse events will be assessed according Common Terminology Criteria of Adverse Events (CTCAE) v.3.0 and analysed as number per patient and number per cycle.
Quality of life | 0,1, 6, 12, 18, 24 months
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of life questionnaire (QLQ) for head and neck cancer patients (HN35) questionnaire filled in by the patients

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Guntinas-Lichius, Prof. Dr., Principal Investigator — Friedrich-Schiller-University Jena
Locations (4):
- Germany (4):
  - Städt. Kliniken Bielefeld gem. GmbH, Bielefeld
  - Friedrich-Schiller-University Jena, Jena
  - Universitätsklinikum Leipzig - Klinik und Poliklinik für HNO-Heilkunde, Leipzig
  - Klinikum Ernst von Bergmann, Potsdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Inhestern J, Schmalenberg H, Dietz A, Rotter N, Maschmeyer G, Jungehulsing M, Grosse-Thie C, Kuhnt T, Gorner M, Sudhoff H, Wittekindt C, Guntinas-Lichius O. A two-arm multicenter phase II trial of one cycle chemoselection split-dose docetaxel, cisplatin and 5-fluorouracil (TPF) induction chemotherapy before two cycles of split TPF followed by curative surgery combined with postoperative radiotherapy in patients with locally advanced oral and oropharyngeal squamous cell cancer (TISOC-1). Ann Oncol. 2017 Aug 1;28(8):1917-1922. doi: 10.1093/annonc/mdx202. PMID 28498880
- [Derived] Inhestern J, Oertel K, Stemmann V, Schmalenberg H, Dietz A, Rotter N, Veit J, Gorner M, Sudhoff H, Junghanss C, Wittekindt C, Pachmann K, Guntinas-Lichius O. Prognostic Role of Circulating Tumor Cells during Induction Chemotherapy Followed by Curative Surgery Combined with Postoperative Radiotherapy in Patients with Locally Advanced Oral and Oropharyngeal Squamous Cell Cancer. PLoS One. 2015 Jul 17;10(7):e0132901. doi: 10.1371/journal.pone.0132901. eCollection 2015. PMID 26186556
- [Derived] Oertel K, Spiegel K, Schmalenberg H, Dietz A, Maschmeyer G, Kuhnt T, Sudhoff H, Wendt TG, Guntinas-Lichius O. Phase I trial of split-dose induction docetaxel, cisplatin, and 5-fluorouracil (TPF) chemotherapy followed by curative surgery combined with postoperative radiotherapy in patients with locally advanced oral and oropharyngeal squamous cell cancer (TISOC-1). BMC Cancer. 2012 Oct 20;12:483. doi: 10.1186/1471-2407-12-483. PMID 23083061